CLINICAL TRIAL: NCT02271555
Title: Inonu University, Turgut Ozal Medical Center, Department of Anesthesiology and Reanimation Malatya
Brief Title: The Effects of Remifentanil on Attenuating the Hemodynamic Responses After Electroconvulsive Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Feray Erdil, Associated professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Inonu 3
Record Dates: First submitted 2014-10-16; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Haemodynamic Rebound
Keywords: electroconvulsive therapy; sevoflurane; remifentanil
MeSH Terms: interventions — Sevoflurane; Remifentanil; Sodium Chloride; Isotonic Solutions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane-remifentanil (Group SR) (Active Comparator): Sevoflurane will be initiated, at 8% for anesthesia induction until loss of consciousness will achieve, at which point it will be discontinued. After the loss of consciousness remifentanil will be administered to Group sevoflurane-remifentanil in the form of a 1 µg/kg intravenous bolus.
  Interventions: Drug: Sevoflurane; Drug: Remifentanil
- sevoflurane-saline (Group SS) (Placebo Comparator): Sevoflurane will be initiated, at 8% for anesthesia induction until loss of consciousness will achieve, at which point it will be discontinued. Placebo is 0.9% saline. After the loss of consciousness saline will be administered to Group sevoflurane-saline in the form of intravenous bolus.
  Interventions: Drug: Sevoflurane; Drug: Saline

INTERVENTIONS:
Drug: Sevoflurane — Anesthetic induction will be achieved via 8% sevoflurane
  Other Names: Sevorane
Drug: Remifentanil — After the loss of consciousness remifentanil will be administered to Group sevoflurane-remifentanil in the form of a 1 µg/kg intravenous bolus.
  Other Names: Ultiva
  Arms: sevoflurane-remifentanil (Group SR)
Drug: Saline — After the loss of consciousness saline will be administered to Group sevoflurane-saline intravenous bolus.
  Other Names: 0.9% isotonic solution
  Arms: sevoflurane-saline (Group SS)

SUMMARY:
The investigators will be evaluated the effects of a single loading dose of remifentanil (1µg/kg), administered as an adjunct to sevoflurane, on duration of hemodynamic profile, seizure activity, and recovery times during electroconvulsive therapy (ECT) in patients with major depression

DETAILED DESCRIPTION:
Major depressive patients will enrolled this trial. Mean arterial pressure (MAP) and heart rate (HR) and peripheral oxygen saturation values will be recorded prior to anesthetic induction (T1); following anesthetic induction (T2); and 0, 1, 3, and 10 minute after the seizure have ended (T3, T4, T5, and T6, respectively). The peak heart rate during the seizure will be recorded from the Electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive patients

Exclusion Criteria:

* younger than 18 years, pregnant, had a history of myocardial infarction in the previous six months, atrial fibrillation or flutter, heart block, unregulated hypertension, cerebrovascular diseases, known drug allergy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The effects of remifentanil on the heart rate after electroconvulsive therapy | 20 minute
  Prior to anesthetic induction (T1); following anesthetic induction (T2); and 0, 1, 3, and 10 minute after the seizure have ended (T3, T4, T5, and T6, respectively).

SECONDARY OUTCOMES:
Seizure duration | 20 minute
  During electroconvulsive therapy
The effects of remifentanil on the mean arterial pressure after electroconvulsive therapy | 20 minute
  Prior to anesthetic induction (T1); following anesthetic induction (T2); and 0, 1, 3, and 10 minute after the seizure have ended (T3, T4, T5, and T6, respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Feray Erdil, MD, Principal Investigator — İnonu Univercity Medical Faculty Department of Anestheisology and Reanimation
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

REFERENCES:
- [Result] Nishikawa K, Higuchi M, Kawagishi T, Shimodate Y, Yamakage M. Effect of divided supplementation of remifentanil on seizure duration and hemodynamic responses during electroconvulsive therapy under propofol anesthesia. J Anesth. 2011 Feb;25(1):29-33. doi: 10.1007/s00540-010-1049-4. Epub 2010 Nov 30. PMID 21116659